CLINICAL TRIAL: NCT00944593
Title: A Randomized Controlled Trial of Gastric Meal With and Without Prior Jejunal Feeding on GI Symptoms and Response in Patients With Diabetic Gastro-enteropathy, Diabetic Controls and Healthy Volunteers
Brief Title: Gastric vs Jejunal Feeding in Diabetic Gastroparesis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Principle Investigator moved to another institution. Research funds transferred. Study to be performed at new institution
Sponsor: University of Zurich (Other)
Collaborators: Schweizerischer Nationalfonds (Other)
Responsible Party: Principal Investigator, MFox, Consultant Gastroenterologist, University of Zurich
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SNF 320030-120597
Record Dates: First submitted 2009-07-20; First posted 2009-07-23 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Diabetic Gastroparesis
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 300kcal liquid Nutrient (Experimental): 300kcal liquid nutrient delivered by NJ tube over 60 minutes before ingestion of a standard oral liquid nutrient test meal
  Interventions: Dietary Supplement: Jejunal Feed
- Normal Saline (Placebo Comparator): Normal Saline delivered via NJ tube over 60 minutes ahead of a standard liquid nutrient test meal
  Interventions: Dietary Supplement: Normal Saline

INTERVENTIONS:
Dietary Supplement: Jejunal Feed — Liquid nutrient (Ensure 200ml (300kcal) over 60 minutes) will be delivered by naso-jejunal feeding tube (previously placed by endoscopy)
  Other Names: Ensure Vanilla, Abbott
  Arms: 300kcal liquid Nutrient
Dietary Supplement: Normal Saline — 200ml Normal Saline 0.9%
  Other Names: Normal Saline 0.9%, Baxter
  Arms: Normal Saline

SUMMARY:
Diabetic 'Gastroparesis' or 'Gastroenteropathy' is a condition in which patients suffer episodes of nausea, vomiting, abdominal bloating and pain after eating. These symptoms occur in the absence of any structural abnormality of the stomach, rather abnormal gastric function underlies the condition. Up to one in five patients with type I diabetes experience symptoms consistent with this diagnosis. The effects on diabetic control, physical health and emotional quality of life are severe. Patients do not respond reliably to general supportive management or conventional medications. Surgical options have disappointing results. The need for more effective treatment is acknowledged universally.

Feeding into the small bowel beyond the stomach (jejunal feeding) is established management in diabetic patients with gastroenteropathy that are malnourished due to poor oral intake. The benefits have been assumed secondary to improved nutrition and diabetic control; however this assertion has never been studied. Recently we observed that patients with severe gastroenteropathy recovered promptly and could eat normally during and for a few hours after jejunal feeding. These observations suggest that jejunal feeding has 'quasi-pharmacological' effects in patients with gastroenteropathy. One attractive explanation for these observations is that gastroenteropathy represents a failure of oral intake to 'switch' the stomach from the fasted to the fed state. According to this hypothesis, jejunal feeding 'restores' the normal fed state by bypassing the dysfunctional stomach.

This project will assess the effects of feeding on gastrointestinal (GI) sensory and motor function in diabetic gastroenteropathy. Healthy volunteers and diabetic controls without symptoms will also be investigated. Studies will assess:

1. Effects on GI symptoms and function to gastric distension in fasted and fed states
2. Effects on GI symptoms and function to oral vs. nasogastric delivery of a test meal
3. A trial of gastric feeding with and without prior jejunal feeding on GI symptoms and function Non-invasive magnetic resonance imaging (MRI) techniques will be applied to assess complex gastric response to feeding. In addition the effects of feeding on symptoms and gastric function will be related to alterations in GI hormones and autonomic nervous activity (eg cardiovagal tone) to assess how the integrated response of the GI tract to feeding fails in patients with diabetic gastroenteropathy.

The primary aim of this project is to assess the effectiveness of jejunal feeding in the management of diabetic gastroenteropathy. However, by defining the processes that 'switch' gastric function between the fasted and the fed states and control gastric emptying, we hope also to identify candidate targets for more effective pharmacologic treatment of this severe disease.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria: • Type 1 diabetes mellitus, confirmed by history of persistent insulin treatment from 12 months' or less after diagnosis, and fasting C peptide concentration of <0.16nmol/L.74

* At least moderate symptoms of gastroenteropathy (GCSI >27)
* Delayed gastric emptying on breath test performed at screening (if no results available)

Disease control

* Type 1 diabetes mellitus, confirmed by history of persistent insulin treatment from 12 months' or less after diagnosis, and fasting C peptide concentration of <0.16nmol/L.74
* Not more than mild symptoms of gastroenteropathy / dyspepsia (GCSI <14).
* Normal gastric emptying on breath test performed at screening (if no results available)

Normal control

* Healthy volunteers recruited by advertisement.
* Not more than mild symptoms of gastroenteropathy / dyspepsia (GCSI <14).
* Normal gastric emptying on breath test performed at screening (if no results available)

General inclusion criteria

* Aged at least 18 and not more than 55 years.
* Body Mass Index: 19-27 kg/m2
* Ability to communicate with the investigator and comply with requirements for entire study.
* Ability to provide written, informed consent

Exclusion criteria: General exclusion criteria

* Gross retention of gastric contents (e.g. bezoar) or evidence of peptic ulcer disease or significant pathology (other than reflux oesophagitis) on upper gastrointestinal endoscopy
* History of gastro-intestinal surgery (except appendicectomy and hernia repair).
* History of abdominal radiotherapy or malignancy
* Mental impairment or psychological disease limiting ability to comply with study requirements
* Progressive or unstable co-morbid condition requiring treatment or precluding safe endoscopic placement of naso-jejunal feeding tube.
* Patients at risk of pregnancy without effective contraception
* Evidence or history of drug or alcohol abuse within two years.
* Unable or unwilling to stop medications influencing upper GI motility

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2011-01

PRIMARY OUTCOMES:
Improvement in symptoms of gastroparesis (GCSI score) | After administration of test meal
  Comparison will be made of symptoms of gastroparesis (GCSI score) after test meal with and without prior jejunal feeding. Symptoms will be assessed after administration and at regular 15 min intervals for 120 min. An integrated score will be calculated.

SECONDARY OUTCOMES:
Gastric emptying rate at gastric emptying half time | 120 min
  A 400ml liquid test meal will be taken. Dynamic change in gastric volume over time will be assessed using a validated 4 parameter model. Gastric emptying rate will be assessed at the time half the gastric volume has left the stomach ("gastric emptying half time")

CONTACTS AND LOCATIONS:
Overall Officials: Innere Medizin: Forschungsgruppe GI-Motility, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland